CLINICAL TRIAL: NCT03851185
Title: Individualised Fluid Management in Haemodialysis: Combining Bioimpedance and Absolute Blood Volume Measurements for Improved Clinical Effectiveness and Patient Experience
Brief Title: Combining Bioimpedance and Blood Volume Measurements in Haemodialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RL18/109517
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Haemodialysis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Around 60,000 patients in the UK are being treated for severe kidney failure. The most common treatment is haemodialysis (HD). An important part of HD is removing extra fluid from the body which the kidneys normally remove in urine. Deciding how much fluid to remove is not easy. It is normally based on clinical signs, such as blood pressure or tissue swollen with fluid, but there is a need for better tests to help guide these decisions.

Bioimpedance tests are one way of measuring fluid status. They involve passing a small electric current through tissue using stickers on the skin. The test is portable, cheap, simple, painless and harmless. One bioimpedance device, the Body Composition Monitor (BCM), has been designed particularly for kidney patients. However the BCM measures fluid in the whole body and cannot tell us how much fluid is in the blood (the blood volume), which has the biggest effect on patients' health.

The aim of this study is to see whether blood volume measurements can help to make fluid management more individualised. This could reduce the impact of dialysis on patients' health and improve patients' experience of the treatment.

Objective 1: To demonstrate whether the addition of blood volume measurements can help to tailor fluid management to HD patients' individual needs. In particular we will look at how body size, nutritional state, age and localised fluid can affect patients' blood volume.

Objective 2: To see if there is a simple way of making blood volume measurements with no need for expertise or extra equipment.

It is planned to recruit 40 patients into 4 clinically different groups and compare results between them.

The results will be compared between groups to help us understand how decisions about fluid management can be tailored to keep blood volume at the optimal level.

ELIGIBILITY:
Cohort 1 - Reference group: This group is intended to represent HD patients who have normal fluid status and normal compartmental fluid volumes.

Inclusion criteria:

* Ultrafiltration volumes in the preceding two weeks of less than 0.5 litres;
* pre-HD BCM-measured OH <1.1 litres; pre-HD blood pressure <140/90.

Cohort 2 - High BMI group: This group is intended to represent patients with high BMI who routinely finish dialysis with significant fluid depletion, as defined by BCM, without intradialytic symptoms.

Inclusion criteria:

* BMI>30 with target weight > 1.1 kg below normally hydrated weight;
* no recorded symptoms related to fluid removal in the preceding 2 weeks.

Cohort 3 - Low LTI group: This group is intended to represent patients who have a low LTI and who routinely finish dialysis with a degree of excess fluid as defined by BCM.

Inclusion criteria:

* LTI < 10kg/m2 with target weight > 1.1 kg above normally hydrated weight.

Cohort 4 - Localised oedema group: This group is intended to represent patients who have localised lower limb oedema.

Inclusion criteria:

* Oedema as defined by pitting

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those receiving haemodialysis
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of post-dialysis blood volume (ABV) in the high BMI group. | 10 mins
  Absolute blood volume measurements: ABV measurements will be made based on the infusion of ultra-pure dialysate into the extracorporeal blood circuit and the analysis of the effect of the dilution on RBV.
Measurement of post-dialysis blood volume (ABV) in the low lean tissue index (LTI) cohort | 10 Mins
  Absolute blood volume measurements: ABV measurements will be made based on the infusion of ultra-pure dialysate into the extracorporeal blood circuit and the analysis of the effect of the dilution on RBV.
Measurement of post-dialysis blood volume (ABV) in the localised oedema cohort | 10 mins
  Absolute blood volume measurements: ABV measurements will be made based on the infusion of ultra-pure dialysate into the extracorporeal blood circuit and the analysis of the effect of the dilution on RBV.

CONTACTS AND LOCATIONS:
Locations (1):
- St James's University Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided